CLINICAL TRIAL: NCT04761172
Title: Near-infrared Fluorescence Imaging With IndoCyanine Green for the Intraoperative Identification of Gastrointestinal Stromal Cell Tumours: a Pilot Study
Brief Title: NIR Fluorescence Imaging With ICG for the Intraoperative Identification of Gastrointestinal Stromal Cell Tumours
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, javanderhage, Prof. dr., Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL67828.058.18
Record Dates: First submitted 2021-01-11; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: GIST

STUDY DESIGN:
Intervention Model Description: Open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Intraoperative near-infrared fluorescence imaging using indocyaninegreen — ICG administration before/during surgery and using near-infrared fluorescence imaging for intra-operative detection and identification of GISTs

SUMMARY:
This is an open-label pilot study including 10 GIST patients scheduled for an elective open or laparoscopic resection at Leiden University Medical Center (LUMC) and Erasmus Medical Center (EMC), Rotterdam. Patients will receive a single dose injection of 10mg ICG at a given moment during the 24 hours prior to surgery or during surgery. The timing of administration will be determined according to a step-up, step-down procedure. Standard of care surgery will be performed and a NIR fluorescence imaging system will be used to record the GIST under fluorescence.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with GIST by histology or cytology, localized or metastasized, scheduled to undergo an elective open or laparoscopic resection.
* 18 years

Exclusion Criteria:

* History of an allergy or hypersensitivity to sodium iodide, iodine or ICG
* Patients with hyperthyroidism and patients with an autonomous thyroid adenoma
* Patients pregnant or breastfeeding
* Patients with severe renal insufficiency (eGFR <30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary tumor detection | Intra-operative
  Tumor detection perceived by the surgeon with and without NIR-imaging

SECONDARY OUTCOMES:
Detection of peritoneal tumor depositions | Intra-operative
  Detection of peritoneal tumor depositions by the surgeon with and without NIR-imaging
Tumor to background ratio | Through study completion, estimated to be 6 months
  Pixel intensity ratio on static images

CONTACTS AND LOCATIONS:
Overall Officials: J. A. van der Hage, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No
On request anonymized data can be shared with other researchers